CLINICAL TRIAL: NCT06645275
Title: Point-of-Care Testing (POCT) for Guided Precision Anticoagulation With Warfarin: A Multicenter, Non-concurrent Controlled Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIT-2024-0271
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Anticoagulation
Keywords: warfarin; POCT; Genetic test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POCT group (Experimental)
  Interventions: Genetic: POCT test
- pyrosequencing group (No Intervention)

INTERVENTIONS:
Genetic: POCT test — Patients undergo POCT testing on the day of warfarin administration, and based on the POCT results, the initial and maintenance doses of warfarin are determined according to the IWPC algorithm.
  Arms: POCT group

SUMMARY:
This study aims to compare the key clinical indicators such as the time to achieve INR target, frequency of dose adjustment, and the incidence of thrombotic and hemorrhagic events between Point-of-Care Testing (POCT) and pyrosequencing technology in the precision dosing of warfarin, in order to assess whether POCT-based warfarin genetic testing is beneficial for improving the quality of anticoagulation treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, gender unrestricted;
* Inpatients in the cardiology department and cardiovascular surgery department who are using warfarin for the first time and require continuous treatment for at least 3 months;
* The patient or legal guardian agrees to the research plan and signs an informed consent form;

Exclusion Criteria:

* Patients with contraindications to anticoagulant therapy or those who are scheduled for surgery in the near future;
* Known genotypes CYP2C9 or VKORC1;
* Patients scheduled to undergo interventional procedures (such as radiofrequency ablation, cardiac defibrillation) in the near future;
* Patients with hematological disorders, bleeding disorders, or a tendency to bleed;
* Patients with severe liver and kidney dysfunction (CrCl < 15ml/min);
* Patients with concurrent tumors, severe immune system diseases, or other terminal diseases;
* Patients with severe heart failure (NYHA Class IV) or severe anemia (hemoglobin < 60g/L);
* Pregnant and lactating women;
* Uncontrolled hypertension (systolic blood pressure > 180mmHg or diastolic blood pressure > 120mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The time it takes for patients to reach the target INR range (INR 2.0-3.0). | Patients will be scheduled for outpatient clinic or phone visits at intervals of 2, 4, 6,13,20,35,60 and 90 day following enrollment.

SECONDARY OUTCOMES:
Percentage of time within the therapeutic range (TTR) | Patients will be scheduled for outpatient clinic or phone visits at intervals of 2, 4, 6,13,20,35,60 and 90 day following enrollment.
Number of warfarin dose adjustments within 90 days | Patients will be scheduled for outpatient clinic or phone visits at intervals of 2, 4, 6,13,20,35,60 and 90 day following enrollment.
Number of times INR is below 2.0 or above 3.0 within 90 days | Patients will be scheduled for outpatient clinic or phone visits at intervals of 2, 4, 6,13,20,35,60 and 90 day following enrollment.
Thrombotic events | Patients will be scheduled for outpatient clinic or phone visits at intervals of 2, 4, 6,13,20,35,60 and 90 day following enrollment.
Cost-effectiveness analysis of POCT and pyrosequencing test | Patients will be scheduled for outpatient clinic or phone visits at intervals of 2, 4, 6,13,20,35,60 and 90 day following enrollment.
bleeding events | Patients will be scheduled for outpatient clinic or phone visits at intervals of 2, 4, 6,13,20,35,60 and 90 day following enrollment.

IPD SHARING:
Plan to Share IPD: No